CLINICAL TRIAL: NCT01491022
Title: A Randomized Trial to Evaluate Ampyra for Gait Impairment in Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Principal Investigator, Corneliu C Luca, Neurology Instructor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110173
Record Dates: First submitted 2011-12-08; First posted 2011-12-13 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Parkinson's Disease
Keywords: parkinson's; gait dysfunction; ampyra; 4-aminopyridine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ampyra (Experimental): Ampyra 10 mg po BID for 4 weeks followed by placebo 4 weeks
  Interventions: Drug: Ampyra first, then Placebo
- Placebo (Sham Comparator): placebo 4 weeks followed by Ampyra 10 mg po BID
  Interventions: Drug: placebo first, then Ampyra

INTERVENTIONS:
Drug: Ampyra first, then Placebo — 10 mg po bid for 4 weeks followed by placebo 4 weeks.
  Other Names: first intervention
  Arms: Ampyra
Drug: placebo first, then Ampyra — placebo
  Other Names: second intervention
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of AMPYRA on a number of symptoms in Parkinson's disease. AMPYRA is a medication approved by FDA for gait dysfunction in multiple sclerosis. There are multiple studies to suggest that persons with multiple sclerosis benefit from this medication and have major improvements in gait after taking this medication. However, this medication was never studied in Parkinson's disease. This study aims to learn about possible benefits of AMPYRA in Parkinson's disease (PD).

DETAILED DESCRIPTION:
Subjects with Parkinson's disease will be randomly assigned to two groups. One group will receive Ampyra first for 4 weeks, followed by 2 weeks break and than 4 weeks placebo while the second group will first receive placebo and then Ampyra.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD with stage Hoehn and Yahr Stage>2-3 and with gait freezing or postural instability.
* On stable dosage dopamine agonist/levodopa, and expected to remain on the same dosage of treatment for the duration of study
* Age less than 80, onset of disease at age more than 45.
* Able to give consent

Exclusion Criteria:

* Past medical history of seizures,
* History of renal insufficiency,
* History of cardiac arrhythmia,
* Severe arthritis,
* Women of childbearing potential,
* Cognitive impairment
* Age more than 80.
* PD patients stage 4 H&Y
* PD patient with recent introduction of dopamine agonist or IMAO B
* PD patients participating in other studies

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corneliu Luca, Study Chair — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Ampyra Then Placebo: Ampyra 10 mg po BID for 4 weeks followed by 2 weeks washout followed by 4 weeks placebo
- Placebo Then Ampyra: placebo for 4 weeks followed by 2 weeks washout followed by 4 weeks Ampyra 10 mg po BID
Period: Intervention 1
Arm/Group | Ampyra Then Placebo | Placebo Then Ampyra
Started | 10 | 12
Completed | 9 | 11
Not Completed | 1 | 1
Period: 2 Week Washout
Arm/Group | Ampyra Then Placebo | Placebo Then Ampyra
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0
Period: Intervention 2
Arm/Group | Ampyra Then Placebo | Placebo Then Ampyra
Started | 9 | 11
Completed | 8 | 11
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Then Ampyra: Placebo for 4 weeks followed by 2 weeks washout followed by Ampyra 10 mg po bid for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Ampyra Then Placebo | Placebo Then Ampyra | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (10.8) | 67.4 (5.9) | 67.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Velocity
Description: The primary outcome measure will be the change in gait velocity as measured with by 3-dimensional gait analysis system.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Ampyra: Ampyra 10 mg po BID
  Dalfampridine: 10 mg po bid for 4 weeks
- Placebo: placebo: placebo
Arm/Group | Ampyra | Placebo
Number analyzed (Participants) | 20 | 20
m/s | 0.03 (0.03) | 0.05 (0.03)

2. Secondary Outcome: United Parkinson's Disease Rating Scale Score(UPDRS) ,
Description: change in UPDRS score (motor) range 0-104, where 0 is good and 104 is worse.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ampyra | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | 35.22 (14.4) | 35.55 (13.7)

3. Secondary Outcome: Freezing of Gait Questionnaire (FOGQ)
Description: change in FOGQ score 0- 16, where 0 is normal, 16 is severely impaired
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ampyra Then Placebo | Placebo Then Ampyra
Number analyzed (Participants) | 20 | 20
units on a scale | 13.16 (4.9) | 13.4 (3.7)

4. Secondary Outcome: Timed Up and Go (TUG) Score
Description: time required to perform TUG.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Ampyra Then Placebo | Placebo Then Ampyra
Number analyzed (Participants) | 20 | 20
seconds | 23.25 (15.4) | 20.6 (15.3)

5. Secondary Outcome: Timed 25-foot Walk Test (T25FW)
Description: time required to perform T25FW.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Ampyra Then Placebo | Placebo Then Ampyra
Number analyzed (Participants) | 20 | 20
seconds | 11.6 (5.0) | 11.8 (6.5)

6. Secondary Outcome: Change in Stride Legth
Description: change in stride length as measured by 3 D capture analysis
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ampyra | Placebo
Number analyzed (Participants) | 20 | 20
meters | -0.01 (0.04) | 0.05 (0.04)

ADVERSE EVENTS:
Time Frame: at 10 weeks
Arm/Group | Ampyra | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 5/22 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ampyra (N=22) | Placebo (N=22)
dizzines (Nervous system disorders) | 4 (4) | 1 (1)
urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
balance worsening (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No